CLINICAL TRIAL: NCT02505022
Title: Role Functioning Changes in New Onset Symptoms
Brief Title: Role Functioning Changes NOS
Status: Terminated | Type: Observational
Why Stopped: Recruitment issues
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Will Cronenwett, MD, Northwestern University
Other Study IDs: STU00201133
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Schizophrenia; Psychotic Disorders; Bipolar Disorder
Keywords: Cognition; Early mental illness; Role functioning
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Mental Disorders | interventions — Drug Therapy; Behavior Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment seeking patients: Patients between 18 and 26 who arrive seeing treatment for new-onset mental health symptoms. They will receive treatment as usual, while being assessed overt he course of one year for changes in role functioning.
  Interventions: Drug: Pharmacotherapy; Behavioral: Behavioral treatment

INTERVENTIONS:
Drug: Pharmacotherapy — Participants may receive pharmacotherapy in the course of treatment-as-usual. This observational study does not influence the type of treatment administered.
Behavioral: Behavioral treatment — Participants may receive behavioral treatment in the course of treatment-as-usual. This observational study does not influence the type of treatment administered.

SUMMARY:
During this study the investigators will 1) collect measures of social cognition and social functioning in adolescents and young adults who are experiencing early symptoms of a major mental disorder; and 2) evaluate the predictive value and utility of a new role functioning assessment measure for individuals experiencing changes in their lives after an index episode of mental illness. This will happen in the context of providing treatment-as-usual to individuals who arrive seeking help with the early phases of mental illness.

DETAILED DESCRIPTION:
The early symptoms of major mental disorders, such as bipolar disorder and schizophrenia, can be non-specific, attenuated, or intermittent. These symptoms nevertheless frequently interfere with an individuals' ability to effectively carry-out multiple aspects of their everyday lives, including social, vocational, and educational functioning. Functional changes may in fact occur before individual symptoms reach the threshold for clinical significance. Relying solely on the emergence of early symptoms of psychopathology can delay treatment or lead to the improper selection of treatments that are not effective. Therefore, measuring changes in real-world functioning that correlate with or predate symptoms may be a useful tool for developing an effective treatment plan.

While psychopharmacology and psychotherapy can improve some symptoms of severe mental illness, much less is known about the mechanisms for improving impairments in social cognition. Importantly social cognition affects not just social functioning, but many critical aspects of real-world functioning. Thus, advancing our understanding of how social cognition and real-world functioning change over time, and their association to changing clinical symptoms, will help improve our understanding of early mental illness, and should inform patient care in new ways. Currently, there are only a limited number of tools available for assessing aspects of real-world functioning as they connect to social cognition. Therefore, the overarching goal of the present study is to conduct a pilot study to develop a new tool that measures functioning and evaluate the relationship between this new tool and measures of social cognition and symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 26 years
2. Individuals seeking treatment for psychiatric symptoms in a clinical care setting
3. Able to provide informed consent (age 18-26)
4. Subjects must consent to a review of the medical records in order to track changes in clinical symptoms
5. Fluent in English

Exclusion Criteria:

1. Adults unable to consent
2. Individuals who have not reached the age of 18
3. Pregnant women
4. Prisoners.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adults with emerging psychopathology. Therefore, all subjects we recruit will be in the age range spanning adolescence and young adulthood, who come to a clinic seeking psychiatric care.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-01; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Correlates between Role Functioning Rating Scale (RFRS), clinical symptoms, and social cognition | 1 year

SECONDARY OUTCOMES:
PONS | 1 year
  Profile of non-verbal sensitivity
TASIT | 1 year
  The Awareness of Social Inference Test
BLERT | 1 year
  Bell-Lysaker Emotion Recognition Task
SFS | 1 year
  Social Functioning Scale
UPSA | 1 year
  UCSD Performance-Based Skills Assessment
EPT | 1 year
  Emotional Perspective-Taking Task
FAP | 1 year
  Facial Affect Perception Task
Informant SLOF | 1 year
  Informant Specific Levels of Functioning Scale; administered to an informant of a participant
SLOF | 1 year
  Specific Levels of Functioning Scale
RFS | 1 year
  Role Functioning Scale
ERS | 1 year
  Emotional Reactivity Scale
ASSIST | 1 year
  Alcohol, Smoking and Substance Involvement Screening Test

CONTACTS AND LOCATIONS:
Overall Officials: Will J Cronenwett, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States